CLINICAL TRIAL: NCT06903585
Title: Non-steroidal Anti-inflammatory Drugs in the Prevention of Bone Pain Flares After Palliative Radiotherapy: A Randomized Controlled Trial
Brief Title: Non Steroidal Anti-inflammatory Drugs in the Prevention of Bone Pain Flares After Palliative Radiotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Lara Hilal, Doctor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIO-2024-0045
Record Dates: First submitted 2025-03-25; First posted 2025-03-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Bone Pain Flare; Bone Metastasis
MeSH Terms: interventions — Naproxen; Anti-Inflammatory Agents, Non-Steroidal; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAID arm (Active Comparator): People in this arm will receive the NSAID naproxen for 5 days, starting from the day they first receive palliative radiotherapy, they will take it as an initial dose of 500mg then as 250mg every 8 hours for a total of 5 days.
  Interventions: Drug: Naproxen (Proxen S); Drug: Esomeprazole 20mg once daily
- Placebo arm (Placebo Comparator): People in this arm will receive placebo pills for 5 days, starting from the day they first receive palliative radiotherapy, they will take a placebo pill every 8 hours for a total of 5 days.
  Interventions: Drug: Placebo; Drug: Esomeprazole 20mg once daily

INTERVENTIONS:
Drug: Naproxen (Proxen S) — Naproxen will be given for 5 days starting from the day subjects first receive palliative radiotherapy, it will be taken as an initial dose of 500mg then as 250mg every 8 hours for a total of 5 days.
  Other Names: NSAIDs
  Arms: NSAID arm
Drug: Placebo — Placebo will be given for 5 days starting from the day subjects first receive palliative radiotherapy, it will be given every 8 hours for a total of 5 days.
  Arms: Placebo arm
Drug: Esomeprazole 20mg once daily — Esomeprazole will be given to all subjects as 20mg once daily starting from the day they start palliative radiotherapy and for a total of 5 days.
  Other Names: PPI; Nexium

SUMMARY:
Solid tumors have the tendency to spread to other organs in around 26% of cases, with many cases involving the bone causing severe bone destruction and pain that reduces patients' quality of life. Palliative radiation therapy is used as a standard of care to decrease cancer-related bone pain, as it has been proven to provide pain relief in many patients, either partially or totally, within only a few weeks. However, some patients experience worsening of bone pain especially within the first 10 days after radiation therapy, this is called bone pain flare, and its incidence is estimated to be around 40%. This pain flare tends to further reduce these patients' quality of life considering their main illness, which necessitates its prevention or alleviation.

Non-Steroidal Anti-inflammatory Drugs (NSAIDs) which are a key component of the World Health Organization (WHO) analgesic options used to alleviate cancer pain have not had a good share of published trials in the prevention of bone pain flares.

In this light the investigators aim to conduct a double-blinded, placebo-controlled randomized controlled trial to investigate the effectiveness of NSAIDs, specifically Proxen, in preventing bone pain flares after palliative radiotherapy, and as a secondary endpoint they will compare the quality of life and side effects experienced by patients in either group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Primary Solid tumor (Any type of solid tumor)
* Painful bone metastases which are otherwise uncomplicated (no fracture and no neurologic symptoms due to nerve impingement or compression)
* Baseline pain score on a numeric rating scale (0-10) of at least 2
* Stable dose and schedule of narcotic medications prescribed

Exclusion Criteria:

* Hematologic malignancy
* Previously irradiated bone
* Current use of steroids
* Current use of NSAIDs which cannot be stopped before randomization
* Contraindications for NSAIDs (hypersensitivity, PUD, prior GI bleed, CKD, HTN, HF, AERD/asthma)
* Contraindications for PPIs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a pain flare within the first 10 days after palliative radiation therapy | From enrollment till 10 days after the start of palliative radiotherapy
  Subjects will be monitored for the occurrence of a pain flare during the first 10 days after the start of their palliative radiotherapy through daily phone calls by the research fellow who will ask the necessary questions to fill out the Brief Pain Inventory questionnaire and compare baseline pain scores to follow-up pain scores. This questionnaire has a minimum score of 0 and maximum score of 110, with higher scores indicating more pain. A pain flare will be considered positive if there is:
  * Two-point increase from baseline on a pain scale from 0-10 with no increase in analgesic medication intake OR
  * At least 25% increase in the intake of analgesic (daily oral morphine) with no decrease in pain scores on a pain scale

SECONDARY OUTCOMES:
Change in quality of life from start of palliative radiotherapy till one month after | From enrollment till 30 days after the start of palliative radiotherapy
  Quality of life scores will be assessed through daily phone calls to the subjects performed by the research fellow who will ask the subjects the necessary questions to fill out the European Organization for Research and Treatment of Cancer Core Questionnaire (EORTC QLQ-BM22) and compare the baseline scores to the recent ones. This questionnaire has a minimum score of 22 and a maximum score of 88, with higher scores indicating greater distress and hence lower quality of life. The phone calls will be daily the first 10 days after start of palliative radiotherapy, and then weekly for a total of 30 days after the start of palliative radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Hilal, MD, Principal Investigator — AUBMC; Bassem Youssef, MD, Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided